CLINICAL TRIAL: NCT03915067
Title: A Phase 2 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex for the Treatment of Platysma Prominence
Brief Title: BOTOX® for the Treatment of Platysma Prominence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1936-201-008
Record Dates: First submitted 2019-03-29; First posted 2019-04-16 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Platysma Prominence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received matching placebo as superficial intramuscular injections administered to the platysma muscle on Day 1.
  Interventions: Drug: Placebo
- BOTOX® Low Dose (Experimental): Participants received BOTOX® Low Dose as superficial intramuscular injections administered to the platysma muscle on Day 1.
  Interventions: Drug: BOTOX® purified neurotoxin complex
- BOTOX® High Dose (Active Comparator): Participants received BOTOX® High Dose as superficial intramuscular injections administered to the platysma muscle on Day 1.
  Interventions: Drug: BOTOX® purified neurotoxin complex

INTERVENTIONS:
Drug: BOTOX® purified neurotoxin complex — BOTOX® superficial intramuscular injections.
  Other Names: Botulinum toxin type A purified neurotoxin complex
  Arms: BOTOX® High Dose; BOTOX® Low Dose
Drug: Placebo — Placebo injections.
  Arms: Placebo

SUMMARY:
To assess the efficacy and safety of BOTOX® in adults with moderate to severe platysma prominence.

ELIGIBILITY:
Inclusion Criteria:

* Female participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period
* A female participant is eligible to participate if she is not pregnant (has a negative urine pregnancy result prior to randomization), not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to follow the studies contraceptive guidance during the treatment and follow-up period through study exit.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this study's protocol

Exclusion Criteria:

* Any medical condition that may put the participant at increased medical risk with exposure to BOTOX®, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function
* Participant has an anticipated need for treatment with botulinum toxin of any serotype for any indication during the study (other than study intervention)
* Anticipated need for surgery or overnight hospitalization during the study
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study
* Females who are pregnant, nursing, or planning a pregnancy during the study
* Known immunization or hypersensitivity to any botulinum toxin serotype
* History of alcohol or drug abuse within 12 months of the study
* Participant has tattoos, jewelry, or clothing that cannot be removed, and that obscure the neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (12):
- United States (7):
  - Skin Care and Laser Physicians of Beverly Hills /ID# 236518, Los Angeles, California
  - Skin Research Institute LLC /ID# 238126, Coral Gables, Florida
  - DeNova Research /ID# 238165, Chicago, Illinois
  - MD Laser Skin & Vein /ID# 234532, Hunt Valley, Maryland
  - The Center for Dermatology Cosmetics & Laser Surgery /ID# 235624, Mount Kisco, New York
  - The Practice of Brian S. Biesman MD PLLC /ID# 234461, Nashville, Tennessee
  - Dallas Plastic Surgery Institute /ID# 236528, Dallas, Texas
- Canada (5):
  - Humphrey Cosmetic Dermatology /ID# 236591, Vancouver, British Columbia
  - Pacific Derm /ID# 238236, Vancouver, British Columbia
  - Dermetics Cosmetic Dermatology /ID# 236899, Burlington, Ontario
  - Sweat Clinics of Canada /ID# 236590, Toronto, Ontario
  - Bertucci MedSpa Inc. /ID# 236523, Woodbridge, Ontario

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Garcia JK, Hopfinger RM, Foley C, Whyte J, Gauthier M, Foster B, Patel V. Development and validation of patient-reported outcome measures for platysma prominence. Curr Med Res Opin. 2025 Jul;41(7):1277-1290. doi: 10.1080/03007995.2025.2537898. Epub 2025 Jul 31. PMID 40704633
- [Derived] Rohrich RJ, Bertucci V, Dayan S, Jones D, Solish N, Rivers JK, Weiss RA, Muhn CY, Harutunian C, Park GS, Shimoga S, Lee E, Tong W. Efficacy and Safety of OnabotulinumtoxinA for the Treatment of Platysma Prominence: A Randomized Phase 2 Dose-Ranging Study. Plast Reconstr Surg. 2025 Jan 1;155(1):79-88. doi: 10.1097/PRS.0000000000011472. Epub 2024 Apr 16. PMID 38640068
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow and all-cause mortality tables are based on all participants randomized on Day 1. Adverse events are reported for safety population, which included all participants who were administered study intervention.
Period: Overall Study
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Started | 57 | 59 | 55
Modified Intent-to-treat (mITT) Population (mITT population included all randomized participants who had at least 1 post-baseline assessment of the primary efficacy parameter, the C-APPS, as described in the protocol.) | 53 | 58 | 53
Safety Population (Safety population included all participants who were administered study intervention.) | 56 | 59 | 54
Completed | 47 | 50 | 49
Not Completed | 10 | 9 | 6
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 3 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0
Not completed — Protocol Deviation | 0 | 0 | 1
Not completed — Covid-19 Related Issues | 2 | 4 | 4
Not completed — Randomized With Incorrect C-APPS | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: mITT population included all randomized participants who had at least 1 post-baseline assessment of the primary efficacy parameter, the C-APPS, as described in the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose | Total
Number analyzed (Participants) | 53 | 58 | 53 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (9.59) | 51.8 (9.16) | 48.6 (10.21) | 50.0 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 54 | 50 | 156
  Male | 1 | 4 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 6 | 17
  Not Hispanic or Latino | 48 | 52 | 47 | 147
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Black or African American | 1 | 0 | 1 | 2
  White | 49 | 56 | 49 | 154
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1-Grade Improvement at Day 14 as Rated by Investigator Using the Clinician Allergan Platysma Prominence Scale (C-APPS)
Description: The investigator evaluated the participant's platysma prominence severity using a 5-grade scale C-APPS at maximum contraction where 1= minimal, and 5= extreme. Higher values indicate worsening condition. Data is reported for participants who achieved at least a 1-grade improvement rated on the C-APPS. Percentages are rounded off to whole number at the nearest decimal. Cochran-Mantel-Haenszel (CMH) chi-squared test was used for analysis.
Time Frame: Day 14
Population: mITT population included all randomized participants who had at least 1 post-baseline assessment of the primary efficacy parameter, the C-APPS, as described in the protocol. Overall number analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 50 | 54 | 51
percentage of participants | 12.0 [3.0 to 21.0] | 77.8 [66.7 to 88.9] | 88.2 [79.4 to 97.1]
Statistical Analysis 1: Comparison: Placebo vs BOTOX® Low Dose; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value derived from CMH model stratified by investigator site and C-APPS at Day 1; Rate Difference = 65.8, 95% CI 2-sided [51.5 to 80.1]
Statistical Analysis 2: Comparison: Placebo vs BOTOX® High Dose; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value derived from CMH model stratified by investigator site and C-APPS at Day 1; Rate Difference = 76.2, 95% CI 2-sided [63.6 to 88.9]

2. Primary Outcome: Number of Participants Who Experienced One or More Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. Treatment-emergent adverse events are defined as any event that began or worsened in severity on or after the first dose of study drug or any AE that was present before the first dose of study intervention, but increased in severity or became serious after the first dose of study intervention.
Time Frame: From the first dose of study drug up to end of study (up to Day 120)
Population: Safety population included all participants who were administered study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 56 | 59 | 54
Participants | 13 | 14 | 14

3. Primary Outcome: Pulse Rate at Baseline
Description: Participants were seated for at least 5 minutes, and pulse was counted over 60 seconds and recorded.
Time Frame: Baseline (Day 1)
Population: Safety population included all participants who were administered study intervention.
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 56 | 59 | 54
beats per minute (beats/min) | 73.0 (10.77) | 74.4 (9.77) | 73.6 (10.66)

4. Primary Outcome: Change From Baseline in Pulse Rate at Day 7
Description: Participants were seated for at least 5 minutes, and pulse was counted over 60 seconds and recorded.
Time Frame: Baseline; Day 7
Population: Safety population included all participants who were administered study intervention. Overall number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 46 | 49 | 46
beats/min | 1.0 (8.19) | -0.5 (6.76) | 1.2 (13.86)

5. Primary Outcome: Change From Baseline in Pulse Rate at Day 14
Description: Participants were seated for at least 5 minutes, and pulse was counted over 60 seconds and recorded.
Time Frame: Baseline; Day 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 50 | 54 | 51
beats/min | 0.4 (8.76) | -1.4 (7.96) | 1.3 (10.49)

6. Primary Outcome: Change From Baseline in Pulse Rate at Day 30
Description: Participants were seated for at least 5 minutes, and pulse was counted over 60 seconds and recorded.
Time Frame: Baseline; Day 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 50 | 53 | 53
beats/min | 0.1 (11.57) | -0.9 (7.09) | -0.5 (10.22)

7. Primary Outcome: Change From Baseline in Pulse Rate at Day 60
Description: Participants were seated for at least 5 minutes, and pulse was counted over 60 seconds and recorded.
Time Frame: Baseline; Day 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 46 | 52 | 51
beats/min | 0.4 (11.14) | 0.3 (8.24) | -2.1 (11.62)

8. Primary Outcome: Change From Baseline in Pulse Rate at Day 90
Description: Participants were seated for at least 5 minutes, and pulse was counted over 60 seconds and recorded.
Time Frame: Baseline; Day 90
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 48 | 53 | 52
beats/min | 1.1 (10.58) | -0.9 (8.76) | 0.0 (9.45)

9. Primary Outcome: Change From Baseline in Pulse Rate at Day 120
Description: Participants were seated for at least 5 minutes, and pulse was counted over 60 seconds and recorded.
Time Frame: Baseline; Day 120
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 47 | 50 | 49
beats/min | 0.5 (12.39) | -0.4 (9.24) | 0.8 (11.77)

10. Primary Outcome: Systolic and Diastolic Blood Pressure (BP) at Baseline
Description: Participants were seated for at least 5 minutes, and systolic and diastolic BP was measured.
Time Frame: Baseline (Day 1)
Population: Safety population included all participants who were administered study intervention.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 56 | 59 | 54
millimeters of mercury (mmHg)
  Systolic Blood Pressure | 116.6 (12.62) | 119.7 (14.96) | 120.4 (13.38)
  Diastolic Blood Pressure | 77.2 (9.11) | 76.6 (9.26) | 77.6 (8.81)

11. Primary Outcome: Change From Baseline in Systolic and Diastolic BP at Day 7
Description: Participants were seated for at least 5 minutes, and systolic and diastolic BP was measured.
Time Frame: Baseline; Day 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 46 | 49 | 46
mmHg
  Systolic BP | 1.2 (11.49) | 1.7 (13.37) | -2.0 (11.14)
  Diastolic BP | -0.5 (6.66) | 0.3 (8.43) | 0.2 (8.57)

12. Primary Outcome: Change From Baseline in Systolic and Diastolic BP at Day 14
Description: Participants were seated for at least 5 minutes, and systolic and diastolic BP was measured.
Time Frame: Baseline; Day 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 50 | 54 | 51
mmHg
  Systolic BP | 0.0 (9.29) | 1.9 (13.27) | -1.7 (10.17)
  Diastolic BP | -1.0 (6.99) | 1.1 (8.69) | -0.5 (7.41)

13. Primary Outcome: Change From Baseline in Systolic and Diastolic BP at Day 30
Description: Participants were seated for at least 5 minutes, and systolic and diastolic BP was measured.
Time Frame: Baseline; Day 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 50 | 53 | 53
mmHg
  Systolic BP | -2.0 (9.25) | -0.7 (13.71) | -2.8 (9.56)
  Diastolic BP | -1.3 (7.46) | 0.6 (8.77) | -0.8 (9.01)

14. Primary Outcome: Change From Baseline in Systolic and Diastolic BP at Day 60
Description: Participants were seated for at least 5 minutes, and systolic and diastolic BP was measured.
Time Frame: Baseline; Day 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 46 | 52 | 51
mmHg
  Systolic BP | -1.2 (9.14) | 2.2 (14.49) | -2.6 (15.00)
  Diastolic BP | -0.4 (6.50) | 1.9 (10.03) | -2.4 (9.80)

15. Primary Outcome: Change From Baseline in Systolic and Diastolic BP at Day 90
Description: Participants were seated for at least 5 minutes, and systolic and diastolic BP was measured.
Time Frame: Baseline; Day 90
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 48 | 53 | 52
mmHg
  Systolic BP | 1.4 (11.40) | -0.3 (11.62) | -2.7 (11.89)
  Diastolic BP | -2.4 (8.52) | 0.6 (7.14) | -3.2 (10.18)

16. Primary Outcome: Change From Baseline in Systolic and Diastolic BP at Day 120
Description: Participants were seated for at least 5 minutes, and systolic and diastolic BP was measured.
Time Frame: Baseline; Day 120
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 47 | 50 | 49
mmHg
  Systolic BP | 0.6 (12.05) | 0.1 (14.11) | -1.3 (10.27)
  Diastolic BP | -0.7 (9.92) | -0.4 (10.43) | -0.5 (9.11)

17. Primary Outcome: Respiratory Rate at Baseline
Description: Participants were seated for at least 5 minutes, and breaths were counted for 30 seconds and multiplied by 2.
Time Frame: Baseline (Day 1)
Population: Safety population included all participants who were administered study intervention.
Measure: Mean (Standard Deviation); unit: breaths per minute (breaths/min)
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 56 | 59 | 54
breaths per minute (breaths/min) | 15.6 (2.53) | 15.5 (2.66) | 15.6 (2.51)

18. Primary Outcome: Change From Baseline in Respiratory Rate at Day 7
Description: Participants were seated for at least 5 minutes, and breaths were counted for 30 seconds and multiplied by 2.
Time Frame: Baseline; Day 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 46 | 49 | 46
breaths/min | -0.1 (1.73) | 0.1 (1.80) | -0.2 (1.65)

19. Primary Outcome: Change From Baseline in Respiratory Rate at Day 14
Description: Participants were seated for at least 5 minutes, and breaths were counted for 30 seconds and multiplied by 2.
Time Frame: Baseline; Day 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 50 | 54 | 51
breaths/min | -0.2 (1.20) | -0.1 (2.05) | 0.0 (1.55)

20. Primary Outcome: Change From Baseline in Respiratory Rate at Day 30
Description: Participants were seated for at least 5 minutes, and breaths were counted for 30 seconds and multiplied by 2.
Time Frame: Baseline; Day 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 50 | 53 | 53
breaths/min | -0.3 (1.70) | 0.5 (1.86) | 0.0 (1.63)

21. Primary Outcome: Change From Baseline in Respiratory Rate at Day 60
Description: Participants were seated for at least 5 minutes, and breaths were counted for 30 seconds and multiplied by 2.
Time Frame: Baseline; Day 60
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 46 | 52 | 51
breaths/min | -0.2 (1.83) | -0.1 (1.69) | 0.2 (1.83)

22. Primary Outcome: Change From Baseline in Respiratory Rate at Day 90
Description: Participants were seated for at least 5 minutes, and breaths were counted for 30 seconds and multiplied by 2.
Time Frame: Baseline; Day 90
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 48 | 53 | 52
breaths/min | -0.3 (1.85) | -0.1 (2.00) | -0.2 (2.04)

23. Primary Outcome: Change From Baseline in Respiratory Rate at Day 120
Description: Participants were seated for at least 5 minutes, and breaths were counted for 30 seconds and multiplied by 2.
Time Frame: Baseline; Day 120
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 47 | 50 | 49
breaths/min | -0.7 (1.71) | -0.2 (2.09) | -0.3 (1.85)

24. Secondary Outcome: Percentage of Participants With at Least a 1-Grade Improvement at Day 14 as Rated by Participant Using the Participant Allergan Platysma Prominence Scale (P-APPS)
Description: The participants evaluated their own Platysma Prominence severity using a 5-grade scale where 1= minimal, and 5= extreme. Higher values indicate worsening conditions. Data is reported for participants who achieved at least a 1-grade improvement rated on the P-APPS. Percentages are rounded off to whole number at the nearest decimal. CMH chi-squared test was used for analysis.
Time Frame: Day 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
Number analyzed (Participants) | 50 | 54 | 51
percentage of participants | 18.0 [7.4 to 28.6] | 75.9 [64.5 to 87.3] | 88.2 [79.4 to 97.1]
Statistical Analysis 1: Comparison: Placebo vs BOTOX® Low Dose; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was derived from CMH model stratified by investigator site and P-APPS at Day 1; Rate Difference = 57.9, 95% CI 2-sided [42.3 to 73.5]
Statistical Analysis 2: Comparison: Placebo vs BOTOX® High Dose; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value derived from CMH model stratified by investigator site and P-APPS at Day 1; Rate Difference = 70.2, 95% CI 2-sided [56.4 to 84.1]

ADVERSE EVENTS:
Time Frame: All cause mortality is reported from enrollment to end of study; median time on follow up was 128.0, 127.0 and 129.0 days for placebo, BOTOX low dose and BOTOX high dose, respectively. TEAEs and SAEs were collected from first dose of study drug until 120 days after last dose of study drug; mean duration on study drug was 1 day for placebo, BOTOX low dose and BOTOX high dose, respectively.
Description: All-cause mortality: All participants randomized on Day 1. Serious and non-serious adverse events: Safety population included all participants who were administered study intervention.
Arm/Group | Placebo | BOTOX® Low Dose | BOTOX® High Dose
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/59 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/56 | 2/59 | 0/54
Other Adverse Events (participants affected / at risk) | 10/56 | 6/59 | 8/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=56) | BOTOX® Low Dose (N=59) | BOTOX® High Dose (N=54)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=56) | BOTOX® Low Dose (N=59) | BOTOX® High Dose (N=54)
INJECTION SITE BRUISING (General disorders) | 4 (4) | 4 (6) | 3 (3)
INJECTION SITE HAEMORRHAGE (General disorders) | 3 (3) | 2 (2) | 1 (2)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT03915067/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT03915067/SAP_001.pdf